CLINICAL TRIAL: NCT05036941
Title: A Cluster Randomized Trial of Two Mask Systems (Acteev™ N95 + Acteev™ Fabric Masks vs. Standard N95 + Fabric Masks During Shifts & in Community) in Preventing Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2) in HCWs
Brief Title: A Trial of Two Mask Systems in Preventing SARS CoV-2 in Healthcare Workers (HCW)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascend Performance Materials (Industry)
Collaborators: Jehangir Clinical Development Centre Pvt. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APM/AM/001
Record Dates: First submitted 2021-08-26; First posted 2021-09-08 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: SARS CoV-2 Infection; Influenza -Like Illness
Keywords: Clinical respiratory illness (CRI)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Acteev™ system (Acteev™ N95 masks YQD8008 during shifts+ Acteev™ fabric masks in community)
  Interventions: Device: Acteev™ Masks
- Arm 2 (Active Comparator): Standard system (standard N95 masks during shifts+ fabric masks in community)
  Interventions: Device: Comparison Masks

INTERVENTIONS:
Device: Acteev™ Masks — Participants will wear the mask on every shift for 8 consecutive weeks. Participants in Arm 1 will be supplied adequate number of Acteev™ N95 masks YQD8008 during 8-hour shift and Acteev™ fabric masks for community use.
  Arms: Arm 1
Device: Comparison Masks — Participants will wear the mask on every shift for 8 consecutive weeks. Participants in Arm 2 will be supplied with adequate number of standard N95 masks during 8-hour shift and fabric mask for community use.
  Arms: Arm 2

SUMMARY:
A cluster randomized trial will be conducted to evaluate the difference between an Acteev™ system (Acteev™ N95 masks YQD8008 during shifts+ Acteev™ fabric masks in community) and a standard system (standard N95 masks during shifts+ fabric masks in community) in preventing Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2)in healthcare workers(HCWs).

DETAILED DESCRIPTION:
This is a maximum 10-week (8-week intervention+2-week follow up) two-armed controlled study to investigate efficacy of Acteev™ system (Acteev™ N95 masks YQD8008 during shifts+ Acteev™ fabric masks in community) compared with standard system (standard N95 masks during shifts+ fabric masks in community) in HCWs working in high-risk hospital wards (ICU, emergency), against the prevention of SARS CoV-2 infection. Prospective HCWs will be identified for the study by the study investigator/study team and be invited for participation in the study. All study procedures will begin only after obtaining written informed consent from the subjects. Subjects will be randomized in one of the two arms mentioned below after meeting all the study eligibility criteria: Arm 1:Acteev™ system (Acteev™ N95 masks YQD8008 during shifts+ Acteev™ fabric masks in community) Arm 2: Standard system (standard N95 masks during shifts+ fabric masks in community).

ELIGIBILITY:
Inclusion Criteria:

* Health care workers and allied health care staff working in COVID wards, COVID ICU, Non COVID ICU (This will include all specialty ICUs in the hospital), Casualty/Emergency, Operation Theatre and Pathology lab of the hospital
* Health care workers and allied health care staff involved in performing high risk procedures like suctioning, intubation, nebulized medications, chest physiotherapy, other aerosol generating procedures and handling pathology samples
* Negative COVID 19 RT-PCR test within last 3 days of screening
* COVID 19 vaccinated or non-vaccinated

Exclusion Criteria:

* Unable or refused to consent
* Current respiratory illness, rhinitis and/or allergy
* Currently participating in any other clinical trial
* Beard or facial hair

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2021-11-13 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
The efficacy of Acteev™ system vs standard system in preventing SARS CoV-2 infection in health care workers | 8 weeks of wearing the masks (with the option of increasing to 12 weeks) with 2 weeks of following up.
  • Number of cases with laboratory-confirmed for viral SARS CoV 2 respiratory infection using RT-PCR with or without two or more respiratory symptoms or one respiratory symptom and/or a systemic symptom

SECONDARY OUTCOMES:
The efficacy of Acteev™ system vs standard system in preventing CRI/ILI infection in healthcare workers | 8 weeks of wearing the masks (with the option of increasing to 12 weeks) with 2 weeks of following up
  • Number of cases with Clinical Respiratory illness defined as two or more respiratory symptoms or one respiratory symptom and/or a systemic symptom along with laboratory-confirmed viral and bacterial respiratory infection other than SARS CoV 2 (Including respiratory syncytial virus (RSV), human metapneumovirus(hMPV), influenza A (H3N2), (H1N1) pdm09, influenza B, parainfluenza viruses 1-4, influenza C, rhinoviruses, severe acute respiratory syndrome (SARS) associated coronavirus (SARS-CoV), coronaviruses 229E, NL63,OC43 and HKU1, adenoviruses and Bacteria like Bordetella pertussis, Bordetella parapertussis, Chlamydia pneumoniae, Mycoplasma pneumoniae)

CONTACTS AND LOCATIONS:
Overall Officials: Raina MacIntyre, MD, Principal Investigator — University of New South Wales, Sydney, AUSTRALIA; Vikram Gopal, PhD, Principal Investigator — Ascend Performance Materials; Yantao Z Hughes, PhD, Principal Investigator — Ascend Performance Materials
Locations (1):
- Jehangir Clinical Development Centre (JCDC) Pvt. Ltd, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacIntyre CR, Seale H, Dung TC, Hien NT, Nga PT, Chughtai AA, Rahman B, Dwyer DE, Wang Q. A cluster randomised trial of cloth masks compared with medical masks in healthcare workers. BMJ Open. 2015 Apr 22;5(4):e006577. doi: 10.1136/bmjopen-2014-006577. PMID 25903751
- [Background] Narayan VV, Iuliano AD, Roguski K, Bhardwaj R, Chadha M, Saha S, Haldar P, Kumar R, Sreenivas V, Kant S, Bresee J, Jain S, Krishnan A. Burden of influenza-associated respiratory and circulatory mortality in India, 2010-2013. J Glob Health. 2020 Jun;10(1):010402. doi: 10.7189/jogh.10.010402. PMID 32373326
- [Background] Chavan RD, Kothari ST, Zunjarrao K, Chowdhary AS. Surveillance of acute respiratory infections in Mumbai during 2011-12. Indian J Med Microbiol. 2015 Jan-Mar;33(1):43-50. doi: 10.4103/0255-0857.148376. PMID 25560001
- [Background] Mudhigeti N, Racherla RG, Mahalakshmi PA, Pamireddy ML, Nallapireddy U, Kante M, Kalawat U. A study of influenza 2017-2018 outbreak in Andhra Pradesh, India. Indian J Med Microbiol. 2018 Oct-Dec;36(4):526-531. doi: 10.4103/ijmm.IJMM_18_272. PMID 30880701
- [Background] Gopal V, Nilsson-Payant BE, French H, et al. Zinc-embedded fabrics inactivate SARS-CoV-2 and influenza A virus. Preprint. bioRxiv. 2020;2020.11.02.365833. Published 2020 Nov 4. doi:10.1101/2020.11.02.365833
- [Background] MacIntyre CR, Wang Q, Cauchemez S, Seale H, Dwyer DE, Yang P, Shi W, Gao Z, Pang X, Zhang Y, Wang X, Duan W, Rahman B, Ferguson N. A cluster randomized clinical trial comparing fit-tested and non-fit-tested N95 respirators to medical masks to prevent respiratory virus infection in health care workers. Influenza Other Respir Viruses. 2011 May;5(3):170-9. doi: 10.1111/j.1750-2659.2011.00198.x. Epub 2011 Jan 27. PMID 21477136